CLINICAL TRIAL: NCT07269873
Title: A Sequential Dose Cohort Pharmacokinetic and Safety Study of Implantable Long-Acting Naltrexone Subcutaneous Pellets With or Without Bupropion Compared to Naltrexone IM Injection (Vivitrol®) in Healthy Normal Volunteers
Brief Title: Safety and PK Study of BICX104 With or Without Bupropion Compared to Vivitrol
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioCorRx Pharmaceuticals Inc (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BICX-25-01b; U01DA059994-01 (NIH)
Record Dates: First submitted 2025-09-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adult Male and Female Volunteers
Keywords: Safety; Pharmacokinetics (PK); Opioid Use Disorder (OUD); Alcohol Use Disorder (AUD); Methamphetamine Use Disorder (MUD); Healthy Normal Volunteers; Naltrexone
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism | interventions — Bupropion; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BICX104 (1 Pellet) (Experimental): 1 naltrexone implantable pellet
  Interventions: Drug: BICX104 naltrexone implantable pellet
- BICX104 (1 Pellet) + bupropion XL 450 mg QD (Experimental): 1 naltrexone implantable pellet + daily oral bupropion extended release 450 mg QD
  Interventions: Drug: BICX104 naltrexone implantable pellet; Drug: Bupropion 150 mg XL
- BICX104 (2 Pellets) + bupropion XL 450 mg QD (Experimental): 2 naltrexone implantable pellets + daily oral bupropion extended release 450 mg QD
  Interventions: Drug: BICX104 naltrexone implantable pellet; Drug: Bupropion 150 mg XL
- Vivitrol q 28 days (Active Comparator): Naltrexone intramuscular injection once every 28 days X 3
  Interventions: Drug: Naltrexone (depot)

INTERVENTIONS:
Drug: BICX104 naltrexone implantable pellet — BICX104 naltrexone implantable pellet
  Arms: BICX104 (1 Pellet); BICX104 (1 Pellet) + bupropion XL 450 mg QD; BICX104 (2 Pellets) + bupropion XL 450 mg QD
Drug: Bupropion 150 mg XL — Extended release bupropion
  Arms: BICX104 (1 Pellet) + bupropion XL 450 mg QD; BICX104 (2 Pellets) + bupropion XL 450 mg QD
Drug: Naltrexone (depot) — Vivitrol naltrexone intramuscular injection
  Arms: Vivitrol q 28 days

SUMMARY:
Naltrexone (NTX), an opioid receptor antagonist, has a longstanding history of safe and effective use for the treatment of addictive disorders. NTX is available in several forms, such as daily oral tablets (Revia®) and sustained release monthly injections (Vivitrol®). BioCorRx Pharmaceuticals is currently developing a subcutaneous implantable pellet drug product, BICX104, which contains NTX base anhydrous (997.5 mg) and can be administered via a minor surgical procedure. BICX104 is anticipated to provide plasma concentrations of ≥ 1 ng/mL NTX for 3 months.

Subjects will be enrolled in 4 sequential cohorts and followed for a total of 196 days, comprising an 84-day treatment period, an 84-day follow-up period, and a 28-day post-treatment follow-up period. While therapeutic levels of naltrexone ( ≥ 1 ng/mL plasma concentration) are expected to be maintained throughout the treatment period, intermittent PK sampling will continue through Day 196, at which all subjects are expected to achieve NTX levels below the level of quantitation (BLQ). Safety parameters include assessment of adverse events, vital signs, laboratory parameters, ECG data, and the Columbia Suicide Severity Rating Scale (C-SSRS), and will continue through the final safety visit at Day 196.

A total of 30 healthy normal volunteers will be enrolled sequentially in the following cohorts, listed in sequence:

1. One BICX104 (1.0 g NTX) implantable pellet (n = 8)
2. One BICX104 implantable pellet with 450 mg QD bupropion XL (n = 8)
3. Two BICX104 implantable pellets with 450 mg QD bupropion XL (n = 8)
4. Three consecutive Vivitrol 380 mg injections Q28 days (n = 6) Enrollment will be stratified by biological sex (50% females and 50% males in each cohort)

Subjects will participate in 18 clinic visits over 31 weeks comprising the 3-week screening period, 12-week treatment period, 12-week follow-up period, and 4-week safety follow-up period.

The test products will be BICX104 implantable pellets (dosage: 1 or 2 implants q. 12 weeks), Bupropion XL (dosage: 450 mg QD)

BICX104 will be supplied to the clinical research site in appropriately labeled closed containers; bupropion XL will be supplied in its standard commercial packaging configuration.

The comparator product will be Vivitrol® IM injection (380 mg NTX) (dosage: 1 injection q. 4 weeks) Vivitrol® will be supplied in its standard commercial packaging configuration.

The study assessments will be as follows:

After all screening assessments and the 24-hour Treatment Initiation Visit, safety and PK assessments will occur on Days 3, 5, 7, 14, 21, 28, 42, 56, 70, 84, 98, 112, 126, 140, 154, and 168. Final safety assessments will occur on Day 196. The Treatment Initiation Visit will involve 1 overnight stay and include PK sampling at pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 12, and 24 hours post-dose, in addition to safety assessments.

Safety assessments will include clinical chemistry, hematology, vital signs, physical exam, ECGs, and administration of the Columbia Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent and to read and understand study documents in English or Spanish
2. Female or male subjects aged 18-65 years old
3. In good health, as determined by the study physician, based on complete medical history, physical examination, vital signs measurement, ECG, and laboratory tests within normal ranges, to permit treatment.
4. Meet subjective and objective measures of being opioid-free prior to study treatment initiation, including negative urine drug screen results at screening and enrollment.
5. BMI of 18.5 to 30.0 kg/m2, inclusive.
6. Must agree to comply with all study requirements and be willing to complete entire study.
7. Persons of childbearing potential agree to use acceptable birth control methods and have periodic urine pregnancy testing done during participation in the study

Exclusion Criteria:

1. Have a history of any psychiatric disorder OR suicidal ideation, behavior, or risk of self-harm as evidenced by endorsement of items 2, 3, 4, or 5 on the C-SSRS
2. Have a history of angle-closure glaucoma
3. Have a history of epilepsy, seizure disorder, or head trauma with neurological sequelae (e.g., loss of consciousness that required hospitalization); current anorexia nervosa or bulimia; or any other conditions that increase seizure risk in the opinion of the study medical clinician
4. Have evidence of second or third degree heart block, atrial fibrillation, atrial flutter, prolongation of the QTc interval (> 450 in males or > 470 in females), or any other finding on the screening ECG that, in the opinion of the study medical clinician, would preclude safe participation in the study
5. Have Stage 2 hypertension as determined by the study medical clinician (e.g., greater than or equal to 160/100 in 2 out of 3 readings during screening)
6. Have any elevated bilirubin test value, or AST, ALT or alkaline phosphatase > 1.5 times the upper limit of normal, per laboratory criteria
7. Have a platelet count <100 x 103/μL; known coagulopathy, or need for anticoagulant therapy during the study
8. Have a known allergy or sensitivity to bupropion, naltrexone, or magnesium stearate, or any topical antiseptics or local anesthetics to be used in the implant procedure.
9. Have taken an investigational drug in another study within 30 days of study consent
10. Have a history of any substance abuse disorder, have been prescribed and taken naltrexone or bupropion within 30 days of study consent, or have been administered Vivitrol® within 60 days of study consent
11. Be receiving ongoing treatment with antidepressants, xanthines (i.e., theophylline and aminophylline), systemic corticosteroids, nelfinavir, efavirenz, chlorpromazine, MAOIs, central nervous system stimulants (e.g., Adderall, Ritalin, etc.), or any medication that, in the judgment of the study medical clinician, could interact adversely with study medications
12. Have a current pattern of alcohol, benzodiazepine, or other sedative hypnotic use which would preclude safe participation in the study as determined by the study medical clinician
13. Require treatment with opioid-containing medications (e.g., opioid analgesics) during the study period
14. Have a surgery planned or scheduled during the study period
15. Are currently in jail, prison or any inpatient overnight facility as required by court of law or have pending legal action or other situation (e.g., unstable living arrangements) that could prevent participation in the study or in any study activities
16. Is prone to skin rashes, keloid scars, or irritation, or has a chronic skin condition or any other condition which might predispose them to adverse reactions to the implant procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Cmax | From enrollment through Day 196 (28 Weeks)
  Maximum plasma concentration for naltrexone and 6-beta-naltrexol
Tmax | From enrollment through Day 196 (28 Weeks)
  Time to reach maximum plasma concentration for naltrexone and 6-beta-naltrexol
AUC | From enrollment through Day 196 (28 Weeks)
  Area under the concentration-time curve for naltrexone and 6-beta-naltrexol
Tlast | From enrollment through Day 196 (28 Weeks)
  Time to reach the last quantifiable plasma concentration for naltrexone and 6-beta-naltrexol
Tlast ≥ 1 ng/mL | From enrollment through Day 196 (28 Weeks)
  Time to reach the last quantifiable plasma concentration that is greater than or equal to 1 ng/mL for naltrexone

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment through Day 196 (28 weeks)
  Incidence and severity of adverse events

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect the confidentiality of study participants.